CLINICAL TRIAL: NCT03172546
Title: Clinical, Biological and Genetic Determinants of Oral Anticoagulants' Activity
Brief Title: Determinants of Oral Anticoagulants' Activity
Acronym: ANTIGOAG
Status: Terminated | Type: Observational
Why Stopped: not sufficiency inclusion
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2014_26; 2015-A01596-43 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-05-24; First posted 2017-06-01 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Anticoagulant
Keywords: direct oral anticoagulant; hemorrhagic complication; thrombotic complication; genetic polymorphisms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anti-IIa users: Determination of predictors of anticoagulant activity in a prospective cohort of patients using oral anti IIa anticoagulant including analysis of PK-PD genetic polymorphisms
  Interventions: Genetic: PK-PD genetic polymorphisms
- Anti-Xa users: Determination of predictors of anticoagulant activity in a prospective cohort of patients using oral anti Xa anticoagulant including analysis of PK-PD genetic polymorphisms
  Interventions: Genetic: PK-PD genetic polymorphisms

INTERVENTIONS:
Genetic: PK-PD genetic polymorphisms — PK-PD genetic polymorphisms analysis in patients receiving either anti-IIa or anti-Xa treatment

SUMMARY:
The primary objective of the present study is to determine the clinical, biological and genetic determinants of the anticoagulant activity in patients treated with either anti-IIa or anti Xa oral anticoagulants.

The secondary objective is to determine the clinical, biological or genetic determinants of hemorrhagic or thrombotic complications during a one year follow-up.

Results will lead to a better prediction of both drug response and risk of complications.

DETAILED DESCRIPTION:
Direct oral anticoagulants are changing clinical practices but a better knowledge of factors that may predict both drug response and risk of complications is need.

Anticoagulant activity is influenced by different factors. Because the biological activity is not easy to measure everywhere, it is important to clearly determine factors that are involved.

A cohort of 550 patients that receive either an anti-IIa or an anti-Xa will be recruited.

The primary objective is to determine clinical, biological and genetic determinants of anticoagulant activity.

This objective will be assessed through a multivariate logistic regression (separately for anti-IIa and anti-Xa) with anticoagulant activity as dependent variable.

Variables that will be included in the statistical model are those known or measured at the entry in the cohort such as :

* Clinical factors : age, sex, weight, dosage and time of the last dose
* Biological factors : serum creatinine level, plasma concentration of the drug
* Genetic polymorphisms :

Factor II and CES1 for anti-IIa drugs Factor X, CYP3, CYP3A4, CYP3A5 and ABCG2 for anti-Xa drugs.

By using the same statistical approach and the same variables, predictive factors of either hemorrhagic or thrombotic events will also be evaluated on the whole cohort. The occurence of hemorrhagic and thrombotic complications will then be assessed through a phone call every 3 months during a one-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient receiving direct oral anticoagulant
* Complete blood count and measure of hemostasis planned
* Patient able to give consent
* Patient with health insurance

Exclusion Criteria:

* Patient not able to consent
* Patient under 18 years old
* Patient refusal
* Patient without health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be composed by all patient receiving a direct oral anticoagulant inside the University Hospital whatever the clinical indication
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Measurement of anticoagulant activity level | Baseline
  Multivariate analysis to determine clinical, biological or genetic predictors of anticoagulant activity level as measured by anti-IIa or anti-Xa activity

SECONDARY OUTCOMES:
Occurence of any hemorrhagic complication | One year follow-up
  Multivariate analysis to determine clinical, biological or genetic predictors of hemorrhagic complications under direct oral anticoagulant
Occurence of any thrombotic complication | One year follow-up
  Multivariate analysis to determine clinical, biological or genetic predictors of thrombotic complications under direct oral anticoagulant

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Deplanque, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- University Hospital, Lille, France

IPD SHARING:
Plan to Share IPD: No